CLINICAL TRIAL: NCT02608138
Title: Iodine Status in Portuguese Children and the Role of Salt Fortification in School Canteens
Acronym: IoGeneration
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Center for Health Technology and Services Research (Other)
Responsible Party: Sponsor
Other Study IDs: 153NU2
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Iodine Status in School Aged Children
Keywords: iodine; urine; children; schools; cognitive performance; salt fortification

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine

GROUPS / COHORTS (1):
- 1: Urinary iodine will be measured at one point in time in school children aged 6-12. A sample of salt used at home and schools will be collected to estimate iodine levels.
  Interventions: Other: Iodine status among portuguese school children

INTERVENTIONS:
Other: Iodine status among portuguese school children

SUMMARY:
It is well known that insufficient iodine intakes impairs the production of thyroid hormones, essential for cognitive development and healthy growth.

Although the World Health Organization (WHO) promotes public health measures for an adequate iodine consumption, it is estimated that one in three school age children remain iodine deficient worldwide. Whereas there is no mandatory iodisation programs in Portugal, young infants are among the most vulnerable to iodine deficiency due to their special requirements.

Therefore, the present study aims to evaluate iodine status in school age Portuguese children (6-12y), compare iodine status in children, cognitive outcomes and thyroid health and monitor the use of iodised salt in school canteens exploring potential implications in children's iodine status.

DETAILED DESCRIPTION:
Iodine is essential for the synthesis of thyroid hormones. Thyroid hormones, especially during periods of increased susceptibility, are crucial for neurodevelopment. Inadequate levels of iodine in the diet may lead to a strong and decisive cognitive impairment which poses a major public health challenge. The World Health Organization prioritized the intake of iodine and recommends the universal enrichment of salt with iodine, so it may reach the general population. In 2013 the Portuguese Department of Education (DGE) issued, as a result of the collaboration with the Portuguese Department of Health (DGS) under the National Program to Promote Healthy Eating a directive introducing the use of iodized salt in school canteens. To ensure the effectiveness and the impact of these policies in Portugal, this project aims to (1) evaluate urinary iodine status in school children (6-12 y), (2) monitor the use of iodized salt in schools, (3) explore potential associations between these parameters. The results of this project will be used to educate food service professionals regarding the use of iodized salt and inform the community about the impact of iodine in health, based on the Norwegian model.

In this study a total of 4800 school aged children will be recruited from approximately 160 schools in the north of Portugal. Parents will be asked to complete the CBCL 6-18, Child Behaviour Checklist and a comprehensive questionnaire which will collect data regarding the child lifestyle and diet. A urine sample will be collected from each participant in school and the Raven's Colored Progressive Matrices will be applied to evaluate children cognitive performance. Anthropometry measurements will be also collected.

ELIGIBILITY:
Inclusion Criteria: School children aged 6 to 12 -

Exclusion Criteria:

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: School aged children (6-12 years)
Sampling Method: Probability Sample
Enrollment: 2018 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Urinary Iodine | One time point collection
Salt Iodine | One time point collection

SECONDARY OUTCOMES:
Cognitive Performance | One time point collection
  Raven's Colored Progressive Matrices
Urinary Creatinine | One time point collection
Height | One time point collection
Weight | One time point collection

CONTACTS AND LOCATIONS:
Overall Officials: Conceição Calhau, PhD, Principal Investigator — CINTESIS, Faculty of Medicine of the University of Porto
Locations (1):
- CINTESIS - Faculty of Medicine of the University of Porto, Porto, Portugal